CLINICAL TRIAL: NCT05076292
Title: Low-dose Glucagon for Prevention of Exercise-Induced Hypoglycemia in People With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 78618; 2021-001342-34 (EudraCT Number)
Record Dates: First submitted 2021-09-29; First posted 2021-10-13 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Type 1 Diabetes; Exercise; Hypoglycemia; Glucagon; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity | interventions — Glucagon-Like Peptide 1; Glucagon; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A randomized, single-blinded, placebo-controlled three-arm cross-over study
Who Masked: Participant
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 150 ug glucagon before exercise (Experimental): 150 ug glucagon will be administered subcutaneously just before exercise and placebo will be administered after exercise.
  Interventions: Drug: GlucaGen
- 2*75 ug glucagon before exercise and after exercise (Experimental): 75 ug glucagon will be administered subcutaneously just before exercise and another 75 ug of glucagon will be administered immediately after exercise.
  Interventions: Drug: GlucaGen
- Saline as placebo (Active Comparator): Saline as placebo will be administered in the same amount as glucagon before and after exercise.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: GlucaGen — 150 ug or 75*2 ug glucagon will be administered subcutaneously to the participants before and after exercise.
  Other Names: Glucagon, GlucaGen®, Novo Nordisk, ATC code H04AA01
  Arms: 150 ug glucagon before exercise; 2*75 ug glucagon before exercise and after exercise
Drug: Saline — Saline will be used as placebo before and after exercise.
  Other Names: ATC-code: Natriumklorid isotonisk "BAUER" B05BB01, V07AB
  Arms: Saline as placebo

SUMMARY:
The primary aim of the study is to compare the efficacy of single-administration low-dose glucagon and split-administration low-dose glucagon to placebo for prevention of exercise-induced hypoglycemia in people with type 1 diabetes using insulin pumps and multiple daily injections (MDI).

The secondary aim is to compare the accuracy of three continuous glucose monitors (CGM) during and after exercise in inpatient and outpatient settings.

DETAILED DESCRIPTION:
A randomized, single-blinded, placebo-controlled three-arm cross-over study will be conducted to assess the study objectives. 22 participants with type 1 diabetes will complete three study visits in random order. At every visit the participants will exercise for 60 min receiving different low doses of glucagon before or before and after exercise compared with placebo.

During the visits and in an outpatient period the participants will have 3 different CGM devices installed and the values will be compared with self-monitored blood glucose values.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* T1D ≥ 2 years
* Use of insulin pump or MDI therapy for ≥ 6 months
* Current use of insulin aspart
* HbA1c ≤ 70mmol/mol (8.5%)
* Body mass index (BMI) ≤ 30 kg/m2
* Performs exercise ≥1 time per week

Exclusion Criteria:

* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period and within 30 days prior to study start
* Professional athletes or highly active individuals ( ≥ 5 hours of exercise per week)
* Known or suspected allergies to glucagon or related products
* History of hypersensitivity or allergic reaction to glucagon or lactose
* Allergy to the patch of the CGM devices
* Patients with pheochromocytoma, insulinoma or gastroparesis
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (methods are considered adequate for study enrollment for females: an intrauterine device, hormonal contraception (birth control pills, implant, patch, vaginal ring or injection), a single partner who is sterile or infertile, or sexual abstinence. Contraception is required throughout the study duration. Sterilized or postmenopausal women (>12 months since last period) are not required to use contraception)
* Inability to understand the individual information and to give informed consent
* Current participation in another clinical trial that, in the judgment of the investigator, will compromise the results of the study or the safety of the subject
* Concomitant medical or psychological conditions identified through review of medical history, physical examination and clinical laboratory analysis that, according to the investigator's assessment, makes the individual unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Incidence rate of hypoglycemia (PG < 3.9 mmol/l) | From 0-180 minutes post-intervention

SECONDARY OUTCOMES:
Percentage of time below range (PG < 3.9) | From 0-180 minutes post-intervention
Percentage of time in range (PG ≥ 3.9 mmol/l and ≤ 10.0 mmol/l) | From 0-180 minutes post-intervention
Time (min) to hypoglycemia (PG < 3.9 mmol/l) | From 0-180 minutes post-intervention
Change in plasma glucose levels | From 0-180 minutes post-intervention
Incidence rate of hyperglycemia (PG > 10 mmol/l) | From 0-180 minutes post-intervention
Nadir plasma glucose concentration | From 0-180 minutes post-intervention
Peak plasma glucose concentration | From 0-180 minutes post-intervention
Incremental peak in plasma glucose concentration | From 0-180 minutes post-intervention
Mean plasma glucose concentration | From 0-180 minutes post-intervention
Plasma glucose Area Under the Curve (AUC) | From 0 to 180 min post-intervention
Percentage of time in hyperglycemia (PG > 10 mmol/l) | From 0-180 minutes post-intervention
Change in visual analogue scale (VAS) for nausea, headache, stomachache, injection site pain and palpitations from intervention (tintervention = 0) to 180 min post-intervention | From 0-180 minutes post-intervention
Mean absolute relative difference (MARD) during the 60-minutes exercise session (using SMBG as the reference value) | During exercise
MARD during the three-day outpatient period (using the 5 daily SMBG as the reference value) | During the three-day outpatient period
MARD during the three-hour inpatient study visit (using YSI as reference value) | During exercise
Rate-of change (ROC) accuracy (using SMBG and YSI as the reference value) | During exercise and during the three-day outpatient period
Point accuracy with the Clarke Error Grid Analysis (CEGA) (using SMBG and YSI as the reference value) | During exercise and during the three-day outpatient period

CONTACTS AND LOCATIONS:
Overall Officials: Sissel B Lundemose, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Sissel Banner Lundemose, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No